CLINICAL TRIAL: NCT06020794
Title: The Efficacy of Leukocyte-poor Platelet Rich Plasma (LPPRP) in the Treatment of Chondromalacia Patella - Randomized Controlled Trial
Brief Title: The Efficacy of LPPRP in the Treatment of Chondromalacia Patella
Acronym: LPPRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kayseri City Hospital (Other Government)
Responsible Party: Principal Investigator, Havva Talay Calıs, Prof. Dr., Kayseri City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KayseriCH
Record Dates: First submitted 2023-08-09; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Chondromalacia Patellae
Keywords: Chondromalacia Patellae; leukocyte-poor platelet-rich plasma; magnetic resonance imaging
MeSH Terms: conditions — Chondromalacia Patellae | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: RANDOMIZED CONTROLLED
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): First group (14 people): 4-weeks home exercise program will be given to control group. The exercise program includes quadriceps isometric exercises (holding for 10 seconds, 20 reps), straight leg raises (20 reps holding for 6 seconds), and semi-squatting exercises (20 reps), hip flexors, hamstring and iliotibial band stretching exercises (20-repetitions), strengthening exercises for hip abductors and adductors (holding for 6 seconds with 20 repetitions). These exercises were said to be performed for 30 minutes, once a day, every day for 4 weeks.
  Interventions: Behavioral: Exercise
- LP-PRP Group (Active Comparator): Second group (14 people): LP-PRP injection and 4-week exercise program will be applied by targeting the suprapatellar bursa. The LP-PRPs to be applied will be obtained by centrifugation of the venous blood taken from the patients by manual methods.
  Interventions: Behavioral: Exercise; Biological: LP-PRP

INTERVENTIONS:
Behavioral: Exercise — quadriceps isometric exercises, straight leg raises, semi-squat exercises, hip flexors, hamstring and iliotibial band stretching exercises, strengthening exercises for hip abductors and adductors
Biological: LP-PRP — The LP-PRPs to be applied will be obtained by centrifugation of the venous blood taken from the patients by manual methods.
  Arms: LP-PRP Group

SUMMARY:
Chondromalacia patella(CP) is a common cause of anterior knee pain in the population under 50 years of age. CP is characterized by softening or varying degrees of damage to the patellar cartilage. The positive effects of leukocyte poor-platelet rich plasma (leukocyte poor-platelet rich plasma, LP-PRP) on cartilage repair and degenerative findings are known. However, there is no randomized controlled study on this subject in CP. The aim of this study is to investigate the effect of LP-PRP on pain, function, walking distance and magnetic resonance imaging (MRI) findings in CP patients.The study is the first to investigate the effect of LP-PRP on cartilage measurement with MRI in Chondromalasia Patella. Patients with anterior knee pain who applied to the physical therapy and rehabilitation outpatient clinic of Kayseri City Hospital, patients with Chondromalacia patella in MRI will be included in the study. A total of 40 patients will be randomized into 2 groups. The exercise program will be applied to both groups as a home program for 4 weeks.

DETAILED DESCRIPTION:
A randomized, prospective, controlled study included 28 patients with MRI stage 2 and above Chondromalasia Patella findings. The patients were randomized into 2 groups, group 1 (the group in which 2 doses of suprapatellar bursa were injected with 2 doses of 3 cc LP-PRP at 1-week intervals and a 4-week home exercise program was given) and group 2 (the control group, the group given a 4-week home exercise program). Patients were tested on the Visual Analogue Scale (VAS) day, night and motion, Western Ontario McMaster Universities Osteoarthritis Index (WOMAC), 6-minute walk test (6MWT) at baseline,1st week, 4th week and 12th week and cartilage thickness, including defective cartilage thickness, and Chondromalasia Patella Outerbridge Staging were evaluated on MRI at baseline and 12th week. WOMAC value was taken as the primary outcome measure and MRI cartilage values were taken as the secondary outcome measure.

Clinic Responsible for Research: Physical Therapy and Rehabilitation Clinic of Kayseri City Hospital

ELIGIBILITY:
Inclusion Criteria:

* Chondromalasia Patella stage 2 and above in MRI requested from patients with chronic pain around the patella, who have increased pain in at least one of the activities that carry loads while the knee is flexed (squatting, stepping, running, jumping, jumping) after physical examination and clinical evaluation
* Patients with VAS 3 and above
* Patients over 18 years of age
* Patients without any deformity in the lower extremity

Exclusion Criteria:

* Coagulopathy and/or thrombocytopenia
* Cardiovascular instability or severe disease condition
* Presence of systemic infection or malignancy
* Pregnancy
* Intra-articular injection in the last 6 months
* Stage 3 and above meniscopathy in MRI
* Evidence or suspicion of rupture of the anterior cruciate ligament on MRI

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-11-04 (Actual)

PRIMARY OUTCOMES:
Western Ontario & McMaster Universities Osteoarthritis Index (WOMAC) | at baseline, 1st week, 4th week and 12th week
  It is a disease-specific measurement for knee and hip osteoarthritis. WOMAC is a personalized index with 5 questions for pain, 2 for stiffness, and 17 questions for questioning daily activities. It has different scores from 0 to 4 (0: none, 1: mild, 2: moderate, 3: severe, 4: very severe). Scale lengths of subheadings; pain=20, stiffness=8, physical function=68. Turkish validation is available . A high score indicates poor health.

SECONDARY OUTCOMES:
MRI cartilage thickness | at baseline and 12th week
  MRI protocol; Proton density (PD-TSE) sagittal, proton density fat suppressed (PD-TSE-FS) coronal, T2W axial and T1W sagittal sequences were taken. Cartilage thickness measurements (millimeter) were measured in the medial and lateral facets where the cartilage was thickest and averaged. In addition, cartilage thickness was measured at the level of the defective area. A low score indicates poor health.
MRI defective cartilage thickness | at baseline and 12th week
  MRI protocol; Proton density (PD-TSE) sagittal, proton density fat suppressed (PD-TSE-FS) coronal, T2W axial and T1W sagittal sequences were taken. Cartilage thickness measurements (millimeter) were measured in the medial and lateral facets where the cartilage was thickest and averaged. In addition, cartilage thickness was measured at the level of the defective area. A low score indicates poor health.
MRI Outerbridge Staging | at baseline and 12th week
  MRI protocol; Proton density (PD-TSE) sagittal, proton density fat suppressed (PD-TSE-FS) coronal, T2W axial and T1W sagittal sequences were taken. The CP stage was performed with the Outerbridge Staging System. According to this staging system, normal cartilage is stage 0; softening or edema without cartilage surface irregularity, stage 1; fragmentation of cartilage, fissure formation or focal defect below 50%, stage 2; Fragmentation, fissure formation or defect in 50% or more cartilage, stage 3; ulceration in the cartilage and exposure of the subchondral bone or increased signal in the exposed subchondral bone were classified as stage 4. A high score indicates poor health.

OTHER OUTCOMES:
Visual analog scale (VAS) | at baseline, 1st week, 4th week and 12th week
  It is used to numerically express the pain felt by the patient. A 100 mm line is drawn and one end is no pain (0), and the other end is unbearable pain (100). The patient is asked to indicate his or her pain state on this line. The distance from the point indicated by the patient to the 0 point indicates the patient's pain. The pain experienced by the patients at rest, during the day and at night in the last 2 weeks was questioned and recorded. A high score indicates poor health.
Six minute walk test | at baseline, 1st week, 4th week and 12th week
  It is a test used to reveal submaximal functional performance. The test should be performed in a closed, quiet environment of at least 30 meters, marked every 3 meters, and in a straight corridor. The patient should be warned to wear comfortable clothes and suitable shoes. The turning points during walking should be marked with the help of a cone and the patient should be asked to go around this cone. The test is terminated by calculating the total distance walked in six minutes.A low score indicates poor health.

CONTACTS AND LOCATIONS:
Overall Officials: Havva Prof. Dr. TALAY ÇALIŞ, Principal Investigator — Health Sciences University, Kayseri City Hospital
Locations (1):
- Health Sciences University, Kayseri Medicine Faculty, Kayseri, Turkey (Türkiye)